CLINICAL TRIAL: NCT06189989
Title: The Effect Of The Care Package Applıed To Babıes Whıch Are Monıtored Wıth Temporary Follow-Up Of The Newborn In The Newborn Intensıve Care Unıt On The Duratıon Of Stay In Non-Invasıve Mechanıcal Ventılatıon And Physıologıcal Parameters
Brief Title: Effect of Care Package on Duration of Stay and Physiological Parameters in Non-invasive Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Esma Şeker, Esma Şeker, Okan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: OkanÜniversitesiEsmaŞeker001
Record Dates: First submitted 2023-12-09; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Care

STUDY DESIGN:
Intervention Model Description: control grup and intervention grup
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In addition to the clinical routine care, the newborn temporary tachypnea care package that we created was applied to the babies in the intervention group. Physiological parameters and blood gas results were recorded.
  Interventions: Behavioral: The group to which a care package was applied in addition to the clinical routine care protocol)
- Control group (No Intervention): Only clinical routine care practices were applied to the babies in the control group. Physiological parameters and blood gas results were recorded.

INTERVENTIONS:
Behavioral: The group to which a care package was applied in addition to the clinical routine care protocol) — Intervention Group:
  * Immediately after the newborn's admission to the intensive care unit, mechanical ventilation mode, physiological parameters, blood gas results and descriptive characteristics of the baby were recorded in the "Data Collection and Daily Monitoring Form".
  * In addition to the routine care practices of the clinic (every 3 hours / 8 times a day), the newborn's temporary tachypnea care package was applied. Postural drainage, percussion and vibration were applied 4 times a day for an average of 10-15 minutes.
  * Mechanical ventilation mode and physiological parameters were recorded one hour after 4 daily maintenance applications.
  * Blood gas parameters were evaluated immediately before and 1 hour after the newborn was separated from mechanical ventilation.
  * Physiological parameters were recorded again 1 hour after the first routine nursing care after the newborn was separated from mechanical ventilation.
  Arms: Intervention Group

SUMMARY:
Temporary tachypnea of the newborn can be improved with minimal respiratory support and nursing care given to babies within the first 72 hours of life. Nursing care practices; It includes pain management, aspiration, moistening and warming of the airways, skin care, nutrition, body temperature regulation, positioning and chest physiotherapy practices.

Physiotherapy practices, when applied in accordance with the criteria, can reduce the newborn's respiratory problems and shorten the hospital stay. Although it has been reported that chest physiotherapy practices have a clinically positive effect on newborns, studies in this field are insufficient.

Nowadays, the concept of care package is frequently used, especially in areas where nursing care is very important, such as intensive care. Implementation of care packages in patient care increases the quality of care by ensuring standardization in the clinic. It also contributes to observing improvements in health practices. The positive results of the use of care packages in their application areas and the lack of care package application in babies monitored with temporary tachypnea of the newborn when the literature was scanned have led to the necessity of conducting studies in this field.

The study was planned as a semi-experimental (non-randomized) control group study to examine the effect of the care package applied to babies monitored with temporary tachypnea of the newborn in the neonatal intensive care unit on the duration of stay in noninvasive mechanical ventilation and physiological parameters.

DETAILED DESCRIPTION:
This study was carried out as a semi-experimental control group study to examine the effect of the care package applied to babies monitored with temporary tachypnea of the newborn in the Neonatal Intensive Care Unit of Istanbul Esenler Gynecology and Children's Hospital, on the duration of stay in noninvasive mechanical ventilation and physiological parameters.

Hypothesis 1 (H1): The care package applied to babies monitored with transient tachypnea of the newborn shortens the duration of stay in noninvasive mechanical ventilation.

Hypothesis 2 (H2): The care package applied to babies monitored with transient tachypnea of the newborn positively affects physiological parameters.

Hypothesis 3 (H3): The care package applied to babies monitored with transient tachypnea of the newborn positively affects blood gas parameters.

The research was conducted in the Neonatal Intensive Care Unit of Esenler Gynecology and Children's Hospital between January 2023 and October 2023.

The sample size was determined by power analysis. The power of the sample in the research was calculated with the G*Power 3.1 program. While the type I error amount was 0.05, the power of the test = 0.85 (α=0.05, 1-β=0.84, effect size: 0.7), the minimal sample size was calculated as 60 newborns (30 newborns in each group). 40 newborns were included in the study. The study was completed by including 40 newborns in the neonatal intervention group (the group in which temporary tachypnea of the newborn care package was applied) and 40 newborns in the control group.

Sample selection criteria; of the newborn;

* Being 36 weeks or above according to gestational age
* Birth weight being 1500 grams and above
* Receive noninvasive mechanical ventilation support
* Feeding via orogastric tube
* Parents' consent for the baby to be included in the study

Exclusion criteria from the sample;

* Those with pneumothorax and suspicion
* Those with cranial bleeding or any suspicion of bleeding
* Babies with congenital anomalies affecting breathing
* Babies who are reconnected to mechanical ventilation after being weaned off noninvasive mechanical ventilation
* Babies with neurological diseases (no neurological problems (hypotonia, hypertonic etc.), no history of convulsions, not using sedative drugs, normal cranial USG,
* Babies with any fractures (clavicle, femur, etc.) were excluded from the sample.

The "Data Collection and Daily Monitoring Form", in which some descriptive characteristics of the baby and physiological parameter measurements were evaluated, was used as a data collection tool. In addition, necessary devices (monitor and sphygmomanometer, stopwatch, thermometer, blood gas device) were used to control physiological parameters.

Care Package for Transient Tachypnea (TTN) Current literature was scanned while determining the parameters included in the care package applied in case of temporary tachypnea of the newborn. Expert opinion was taken for the content of the care package prepared in line with the literature (2 academic nurses, 2 clinical nurses and 1 specialist physician). Care Package consists of 5 items.

1. Heating and humidifying the oxygen-air mixture given to the baby
2. Stopping the baby's feeding and switching to open drainage with orogastric tube (OGS)
3. Application of postural drainage, percussion and vibration 4 times a day for an average of 10-15 minutes
4. If necessary, aspirate the baby
5. Changing the position given to the baby (to increase oxygenation) periodically (every 3 hours)

The newborns included in the study were divided into two groups: intervention and control groups. Between the dates of the research, the first 40 newborns who met the sampling criteria were included in the control group (who received nursing care in line with the routine care protocol of the clinic), and the 40 newborns who met the sample criteria (who received nursing care in line with the routine care protocol of the clinic) were included in the control group, and the 40 newborns who met the sample criteria were given training on the care package after the nurses working in the clinic. (in addition to the maintenance package application) were included in the intervention group.

To prevent the research groups from being influenced by each other, the study started with the control group first. Nursing care was applied to the control group in line with the routine care protocol of the clinic. After the control group data were collected, all nurses working in the clinic were given training on the application of the neonatal temporary tachypnea care package to be applied to the intervention group. The training was given within the scope of a presentation prepared by the researcher in the staff room within the clinic. The training was planned according to the nurses' working hours and was planned in 5 separate groups according to the day they were in the hospital and their available hours. The training lasted approximately 20 minutes. After the training was completed, care package applications for the intervention group started.

A data collection and daily monitoring form was filled out for newborns in both groups immediately after admission to the intensive care unit. The newborn was placed in a pre-heated incubator and monitored. A hydrocolloid strip tape was cut and pasted in a T shape on his nose and he was connected to the mechanical ventilator via a ram cannula interface. An oragastric catheter was inserted into the stomach (with a 10ml syringe) and open drainage was performed. Blood samples requested by the physician were taken and a vascular access was established. The patient's intravenous fluid was started. After the newborn was stabilized, care practices were performed every three hours in line with the clinical routine care protocol. Neonatal temporary tachypnea care package was applied to the newborns in the intervention group in addition to the clinical routine until they were weaned from mechanical ventilation support.

Evaluation of Data The data were evaluated with appropriate statistical analysis in the SPSS 21.0 program. Number, percentage, mean and standard deviation were used as descriptive statistical methods in the evaluation of the data. Frequency and percentage distributions of the data are given. In the study, intra-group measurements were made with correlated sample one-way analysis of variance, and inter-group measurements were made with independent group t test. Bonferonni test was applied to determine which group caused the difference. 0.05 was used as the significance level, and if p<0.05 it was stated that there was a significant difference, and if p>0.05 it was stated that there was no significant difference.

ELIGIBILITY:
Inclusion Criteria:

-Being 36 weeks or above according to gestational age

* Birth weight being 1500 grams and above
* Receive noninvasive mechanical ventilation support
* Feeding via orogastric tube
* Parents' consent for the baby to be included in the study

Exclusion Criteria:

* Those with pneumothorax and suspicion
* Those with cranial bleeding or any suspicion of bleeding
* Babies with congenital anomalies affecting breathing
* Babies who are reconnected to mechanical ventilation after being weaned off noninvasive mechanical ventilation
* Babies with neurological diseases (no neurological problems (hypotonia, hypertonic etc.), no history of convulsions, not using sedative drugs, normal cranial USG,
* Babies with any fractures (clavicle, femur, etc.) were excluded from the sample.

Ages: 36 Weeks to 41 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Heart rate Vital Signs | It was evaluated upon admission to intensive care, 1 hour after the first care, and 1 hour after the first care after weaning from mechanical ventilation.
  Heart rate (beats/minute) were evaluated
Respiratory Rate Vital Signs | It was evaluated upon admission to intensive care, 1 hour after the first care, and 1 hour after the first care after weaning from mechanical ventilation.
  Respiratory Rate (breaths/minute) were evaluated
Body temperature Vital Signs | It was evaluated upon admission to intensive care, 1 hour after the first care, and 1 hour after the first care after weaning from mechanical ventilation.
  Body temperature (°C) were evaluated
Oxygen saturation Vital Signs | It was evaluated upon admission to intensive care, 1 hour after the first care, and 1 hour after the first care after weaning from mechanical ventilation.
  Oxygen saturation (%) were evaluated
Blood pressure Vital Signs | It was evaluated upon admission to intensive care, 1 hour after the first care, and 1 hour after the first care after weaning from mechanical ventilation.
  Blood pressure (mmHg) were evaluated
blood gas pH value : | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas H iyon
blood gas PCO2 value | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas PCO2 (mmHg) were evaluted
blood gas HCO3 value | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas HCO3 (mEq/L) were evaluted
blood gas PaO2 value | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas PaO2 (mmHg)were evaluted
blood gas SaO2 value : | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas SaO2 (mmHg)were evaluted
blood gas lactat value | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas lactat (mmol/L) were evaluted
blood gas BE value | It was evaluated upon admission to the intensive care unit, immediately before weaning from mechanical ventilation, and 1 hour after weaning from mechanical ventilation.
  blood gas BE(mmol/L) were evaluted

SECONDARY OUTCOMES:
Total duration of mechanical ventilation stay | 1 hour after discharge from intensive care
  in total hours
Total duration of stay in intensive care unit duration of transition to oral feeding were evaluated). | 1 hour after discharge from intensive care
  in total hours
Total duration of transition to oral feeding were | 1 hour after discharge from intensive care
  in total hours

CONTACTS AND LOCATIONS:
Overall Officials: Gülzade Uysal, Assoc. Dr, Study Director — Okan Üniversitesi
Locations (1):
- Esma Şeker, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No